CLINICAL TRIAL: NCT07374341
Title: The Effectiveness of Guided Botulinum Toxin "A" Injection to the Masticatory Muscles in the Management of Condylar and Subcondylar Fractures (Randomized Controlled Clinical Trial)
Brief Title: The Effectiveness of Guided Botulinum Toxin "A" Injection to the Masticatory Muscles in the Management of Condylar and Subcondylar Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakinam Gheeta (Other)
Responsible Party: Sponsor-Investigator, Pakinam Gheeta, Instructor of oral surgery, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9239261
Record Dates: First submitted 2026-01-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Condylar Fractures; Subcondylar Fracture
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided Botulinum Toxin injection + closed reduction and intermaxillary fixation (Experimental)
  Interventions: Other: BOTOX Cosmetic®; Procedure: Closed reduction and intermaxillary fixation
- Conventional treatment (Active Comparator)
  Interventions: Procedure: Closed reduction and intermaxillary fixation

INTERVENTIONS:
Other: BOTOX Cosmetic® — The BTX vile is diluted with 2.0 cc saline or distilled water. It is 5 BU (Botox) per 0.1cc, so it is easy to measure (for 2.5 cc normal saline, you can calculate as 4 BU per 0.1 cc) therefore, the investigators can easily adjust the amount to be injected into the muscles of Mastication. Using a 5 cc syringe, draw more than 3 cc of air and inject into the botulinum toxin vial. Check whether the air is sucked into the vial. If air is not sucked into the vial, the vial is discarded as the vacuum is not present in the vial, thus it is faulty. To achieve a desirable concentration of dilution solution, an injection of 2.5 cc of normal saline into botulinum toxin and then it is gently mixed. Two to Three days prior to the surgical intervention, the BTX will be injected to the muscles of mastication; the lateral pterygoid, the masseter and temporal is of the fractured site. The, closed reduction and intermaxillary fixation will be performed for fracture management.
  Arms: Ultrasound-guided Botulinum Toxin injection + closed reduction and intermaxillary fixation
Procedure: Closed reduction and intermaxillary fixation — All patients will be treated using the closed reduction and intermaxillary fixation method. The patients will be treated under local or general anesthesia depending on the availability of other concomitant fractures and general status of the patient.

SUMMARY:
The aim of this study, is to evaluate the effectiveness of ultrasound guided injection of botulinum toxin A into the muscles of mastication; the masseter, temporalis and the lateral pterygoid, in a closed reduction approach of condylar and sub-condylar fractures, seeking to shed light on the efficacy and potential advantages of this innovative therapeutic avenue.

ELIGIBILITY:
Inclusion Criteria:

* Having unilateral extra-capsular condylar/ sub-condylar fractures isolated or associated with other fractures.
* Isolated intra-capsular fractures.
* Moderate condylar displacement, JO to 45 degrees or incomplete fractures.
* Reproducible occlusion without drop-back or with drop-back that returns to midline on release of posterior force.
* Availability of more than half of the dentition

Exclusion Criteria:

* Bilateral condylar fractures
* Gross condylar displacement> 45 degrees (severely displaced)
* Anatomic reduction of ramus height 2: 2 mm
* Unstable occlusion (e.g., periodontal disease, less than three teeth per quadrant)
* Patients with severe polytraumas.
* Patients with relative contraindications to BTX injections that may include; pregnancy, lactation, BTX Allergies and presence of infection at the injection site.
* Patients with motor neuron diseases.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | up to 2 weeks
  Will be assessed through a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Occlusion Assessment | up to 3 months
  Assessment of the Occlusion will be performed and given a score:
  1. Same to pre-traumatic
  2. Minor difference
  3. Functional malocclusion
  4. Needs occlusal correction
  5. Gross malocclusion.
Mouth opening | up to 3 months
  Inter-incisal distance will be measured in (cm) using a ruler, to assess the degree of mouth opening.
Mouth deviation assessment | up to 3 months
  The status of the deviation preoperatively, for the example the availability of cross bites or minor deviations, will be compared to the statues three months postoperatively. Photographs will be obtained for all patients to document occlusion and mouth opening.
Time frame needed until the intermaxillary fixation (IMF) is removed | through study completion, an average of 6 months
  The Intermaxillary fixation will be removed once satisfactory occlusion was achieved and time frame of the IMF will be recorded for each patient.
Bone density at the fracture line | 6 months
  An immediate postoperative CT will be obtained, followed by another one taken after 6 months postoperatively. The mean bone density at the fracture line in the 6 months CT-scan will be compared with the immediate postoperative and the preoperative scans and the mean difference between the scans will be calculated.
The angle between fracture and the longitudinal axis of the ramus | 6 months
  An immediate postoperative CT will be obtained, followed by another one taken after 6 months postoperatively. The angle between the condylar or subcondylar fracture, and the longitudinal axis of the ramus will be measured and compared pre-operatively and six months post operatively and the difference will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No